CLINICAL TRIAL: NCT03035266
Title: The Effect of Blood Flow Restriction Training on Muscle Atrophy Following Knee Surgery; A Randomized Control Trial
Brief Title: The Effect of Blood Flow Restriction Training on Muscle Atrophy Following Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Mason, Assistant Chief, PT, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16KACH016
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Knee Injuries
Keywords: blood flow restriction; strength; muscle atrophy; post-operative therapy; knee
MeSH Terms: conditions — Knee Injuries; Muscular Atrophy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized control trial. After consenting, subjects will be randomized to one of two groups by using a computer generated random number.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators recording thigh girth and isokinetic data will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restriction (BFR) (Experimental): All subjects will perform traditional post-operative rehabilitation until discharge from the hospital following surgery and continue until formal discharge from physical therapy upon completion of rehabilitation. One week following surgery, subjects randomized to the BFR group will begin combining BFR with all lower extremity strengthening exercises supervised in clinic up to 3 times per week for 12 weeks.
  Interventions: Other: Blood Flow Restriction
- Standard rehabilitation (control group) (Active Comparator): All subjects will perform traditional post-operative rehabilitation until discharge from the hospital following surgery and continue until formal discharge from physical therapy upon completion of rehabilitation.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: Blood Flow Restriction — Delfi's Personalized Tourniquet System for Blood Flow Restriction has been specifically designed to safely regulate and control tourniquet pressure. Occlusion pressures will be set at 80% of total occlusive pressure as determined by the Doppler sensor. Each subject will perform 4 sets of each exercise (1 set of 30 repetitions followed by 3 sets of 15 repetitions). The pressure will remain through completion of the final set, but not to exceed 5 minutes. One minute rest without tourniquet application will be performed between 5 minute cycles. Sets and repetitions will remain constant for each subject; however, resistance will be incrementally increased after the subject is able to complete all 75 repetitions without loss of proper form.
  Arms: Blood Flow Restriction (BFR)
Other: Standard rehabilitation — Standard of care for post-operative condition
  Arms: Standard rehabilitation (control group)

SUMMARY:
The investigators will compare differences in quadriceps strength, leg girth, and functional outcome scores between two groups of patients after weeks 6 and 12 as well as 6 months following meniscus or articular cartilage repair/restoration requiring 6 weeks of non-weight bearing or limited weight bearing status in a brace at 0° degrees of knee extension. One group will receive BFR with standard post-operative rehabilitation for 12 weeks followed by the standard protocol progression for the remainder of the treatment program. The other group will receive standard post-operative rehabilitation without BFR for the duration of treatment program.

DETAILED DESCRIPTION:
The aim is to compare strength, patient reported outcomes, and functional outcomes of post-operative therapy with and without adjunctive BFR training. To accomplish this task the investigators will compare differences in thigh girth between two groups of patients after the first 6 weeks and 12 weeks as well as 6 months following meniscus or articular cartilage repair requiring 6 weeks of non-weight bearing or limited weight bearing status in a brace at 0˚ degrees of extension. In addition, isokinetic testing of the quadriceps and hamstrings will be performed at 12 weeks and 6 months post-operatively. Lower extremity girth measurements after knee surgery can be performed with good to excellent intra- and inter-rater reliability. Quadriceps strength measured with isokinetic testing is related to performance measures such as jumping. Limb circumference measurement, limb CSA measurement, and isokinetic strength testing are commonly utilized in BFR studies as outcome measures.One group will receive BFR for 12 weeks in addition to standard post-operative rehabilitation and the other group will receive standard post-operative rehabilitation without BFR.

ELIGIBILITY:
Inclusion Criteria:

* Military healthcare beneficiaries between the age of 18 and 50 years.
* Must intend to remain on station at location of surgery for 6 months from date of surgery.
* Meniscus repair or cartilage restoration technique to include microfracture, osteochondral autograft transfer system, osteochondral allograft transplantation, and autologous chondrocyte implantation following standard post-operative protocol guidelines requiring a 6 week period of non-weight bearing or limited weight bearing in a brace at 0˚ degrees of extension.

Exclusion Criteria:

* Concomitant ligamentous repair/reconstruction
* Known pregnancy
* Any medical condition for which aerobic exercise is contraindicated
* Additional back, hip, or knee surgery in the previous 12 months
* History of vascular or cardiac impairment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Peak Torque (foot-pounds), best repetition out of 15 repetitions | 12 weeks and 6 months post operative
  Change in isokinetic peak torque knee extension and knee flexion at 180 degrees/sec and at 300 degrees/second

SECONDARY OUTCOMES:
Thigh circumference (centimeters) | baseline, 6 weeks, 12 weeks, and 6 months
  Change in girth measurements of thigh:
  10 cm from proximal patella 15 cm from proximal patella 33% length from proximal patella to inguinal crease
Visual Analog Scale (VAS), 0 to 40 mm self report pain scale | baseline, 6 weeks, 12 weeks, and 6 months
  Change in VAS for Pain
Lower Extremity Functional Scale (LEFS) Questionnaire | baseline, 6 weeks, 12 weeks, and 6 months
  Change in LEFS Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: John S Mason, DSc, DPT, Principal Investigator — Keller Army Community Hospital
Locations (2):
- United States (2):
  - Keller Army Community Hospital, West Point, New York
  - Womack Army Medical Center, Fort Bragg, North Carolina

IPD SHARING:
Plan to Share IPD: No